CLINICAL TRIAL: NCT05700864
Title: Assessing the Efficacy of Recombinant Human Nerve Growth Factor (rhNGF) Treatment in Patients With Neuropathic Corneal Pain (NCP)
Brief Title: NGF Treatment for Patients With Neuropathic Corneal Pain
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding of study was withdrawn
Sponsor: Tufts Medical Center (Other)
Collaborators: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002840
Record Dates: First submitted 2022-09-06; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Corneal Disease; Neuropathy
MeSH Terms: conditions — Corneal Diseases | interventions — cenegermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oxervate® (cenegermin) (Experimental): OXERVATE™ 0.002% (20 mcg/mL) cenegermin-bkbj
  Interventions: Drug: Cenegermin-Bkbj

INTERVENTIONS:
Drug: Cenegermin-Bkbj — Cenegermin-bkbj ophthalmic solution administered as one drop in both eyes every 3 hours 4 times daily for 4 weeks
  Other Names: OXERVATE™ 0.002% (20 mcg/mL) cenegermin-bkbj ophthalmic solution

SUMMARY:
This prospective, single center, interventional, open-label, single arm, non-randomized trial seeks to investigate the efficacy of Oxervate® (cenergermin 0.002% eye drops) on ameliorating the signs and symptoms of neuropathic corneal pain (NCP). The study aims to enroll 28 subjects with NCP. All patients will be evaluated for clinical symptoms and signs of NCP, corneal staining and nerve regeneration (by IVCM) at Baseline (Visit 2) through the end of study (16 weeks post treatment).

DETAILED DESCRIPTION:
During the screening (Visit 1 / Day -8) all procedures for inclusion will be performed. From the day of screening the participants will stop any kind of further previous ocular treatment regime, except commercially available preservative free artificial tears provided by Sponsor for 7 days and 9 days as maximum (day -8 to day -1+2) until the baseline(Visit 2) . At the end of the washout period (day -8 to day -1+2), participants meeting the entry criteria for this study will be assigned to receive the Oxervate® at 4times/daily dosing in both eyes for 4 weeks.

At Week 1, participants will be queried for adverse events. If the participant reports side effects while on 4times/daily dosing, subjects will be instructed to begin a modified dosing regimen: 4 times daily for 3 days, then 1 day off dosing. At Week 4, participants will be evaluated for clinically significant changes. If resolution of NCP or improvement is observed, Oxervate® will be discontinued. If there is partial/no-improvement, participants will be instructed to begin an increased dosing regimen of 6times/daily. If at any point during the intervention period ocular pain/irritation is worsened for a prolonged period, Oxervate® intervention will be discontinued.

During the 8 weeks of intervention, only the administration of Oxervate® is allowed. Nevertheless, if strictly needed, the participant can take preservative free artificial tears (provided by Sponsor). The use (n° drops/day) of preservative free artificial tears will be clearly documented in a participant's diary and in the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* Symptoms of neuropathic corneal pain at least 3 months, such as burning, stinging, light sensitivity, discomfort or pain.
* Positive ICVM findings
* If female with childbearing potential, have a negative pregnancy test
* Best corrected distance visual acuity, using corrective lenses if necessary, in the study eye of at least +1.0 Log MAR (Snellen <20/200)
* Satisfying all Informed Consent requirements
* Ability and willingness to comply with study procedures
* Ability to speak and understand the English language sufficiently to understand the study, provide written consent, and allow completion of all study assessments

Exclusion Criteria:

* Evidence of any active ocular infection
* Evidence of any intraocular inflammation
* Evidence of any persistent epithelial defect/ulcer
* Evidence of any corneal scar/corneal edema
* Presence of any other ocular conditions that require topical medications
* History of severe systemic allergy or severe ocular allergy
* Inability to suspend topical medications during the duration of the study
* Inability to suspend oral medications for NCP.
* No changes in VAS score after topical 0.5% proparacaine hydrochloride (Alcaine, Alcon, Fort Worth, TX)
* History of any ocular surgery within three months before study Visit 1(day 0)
* Ocular surgery expected during the 16 weeks of the trial
* Use of refractive/therapeutic contact lenses during the study period
* Female patients that are pregnant/have a positive pregnancy test result/are breast-feeding/intend to become pregnant during the study treatment period
* Drug addiction/alcohol abuse within the last year
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of OXERVATE 0.002% 4 times/daily on neuropathic corneal pain as assessed by corneal nerve regeneration. | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  Quantifying total number of nerves of the corneal subbasal nerve plexus through in vivo confocal microscopy IVCM), summation of main trunk and branch nerves in one image reported as frame/nerve. Change from baseline in nerve quantity on IVCM at 16 weeks.
Efficacy of OXERVATE 0.002% 4 times/daily on neuropathic corneal pain as assessed by changes in ocular inflammation on in vivo confocal microscopy | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  Change in dendritic cell density on in vivo confocal microscopy from baseline to 16 weeks. The total nerve density will be assessed as the total nerve length in micrometers per image frame area (0.16mm^2), from the three best representative images of each eye.
Efficacy of OXERVATE 0.002% 4 times/daily on neuropathic corneal pain as assessed by changes in ocular redness using the McMonnies/Chapman-Davies (MC-D) grading scale. | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  Changes in grade of conjunctival hyperemia and bulbar conjunctival redness using the McMonnies/Chapman-Davies (MC-D) scale 0-1-2-3-4-5, 0 being absent conjunctival redness and 5 being severe conjunctival hyperemia

SECONDARY OUTCOMES:
Occurrence of treatment-related adverse events assessed by severity and temporal relationship of study treatment. | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  The severity of each adverse event observed will be evaluated as serious or not serious. Occurrence will be evaluated as expected or unexpected in relation to treatment. The relationship of the event to the study treatment will be assessed by the investigator as possibly, probably, or definitely related.
Tolerability of OXERVATE 0.002% on neuropathic corneal pain as assessed by the ocular surface disease index (OSDI) questionnaire, change from baseline ocular symptom score on OSDI | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  The ocular surface disease index (OSDI) questionnaire is a 12-item assessment of ocular symptoms and their impact on vision-related functioning. Each of the 12 items of the OSDI are graded on a scale of 0 to 4, where 0 indicates none of the time; 1 some of the time; 2 half of the time; 3, most of the time; and 4 all of the time. The total OSDI score is then calculated by the sum of scores for all questions answered, multiplied by 100. This integer is then divided by [total number of questions answered) x 4]. The highest possible score on OSDI questionnaire being 100, represents most severe symptoms, whereas lower OSDI score represent lower symptom severity.
Patient Reported outcome on quality of life dimensions of OXERVATE 0.002% on neuropathic corneal pain as assessed by Ocular Pain Assessment Survey (OPAS), change from baseline ocular pain score on OPAS | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  The Ocular Pain Assessment Survey (OPAS) is a 27-item quantitative questionnaire designed to provide an assessment of the symptoms and quality of life effect of ocular pain. Each of the 27 items is graded on a scale of 0-10, or a scale of 0% to 100%, where 0 indicates none and 10 or 100 indicate maximum. The OPAS questionnaire assess quality of life dimensions by addressing ocular pain intensity, interference with daily activities, aggravating factors and associated symptoms, as well as non-ocular pain. Higher scores indicate greater impact on quality of life, whereas lower scores indicate less interference on quality of life dimensions.
Changes in corneal nerve function as assessed by hyperosmolar eye-drop test, change from baseline pain score on the Visual Analog Scale (VAS) at 16 weeks. | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  Pain score on the Visual Analog Scale graded from 0 to 10, where 0 is no pain and 10 is the worst pain one can imagine before and after a topical drop of hyperosmolar solution is applied to both eyes.
Resolution of peripheral pain component as assessed by proparacaine eye-drop test, change from baseline pain score on the Visual Analog Scale (VAS) at 16 weeks. | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  Pain score on the Visual Analog Scale graded from 0 to 10, where 0 is no pain and 10 is the worst pain one can imagine before and after a topical anesthetic drop (proparacaine) is applied to both eyes. Peripheral pain will be assessed by percent decrease in pain VAS score after topical proparacaine eye drop. Partial (greater than or equal to 50% decrease in pain VAS) or total pain relief with anesthetic drop is indicative of peripheral pain and no response to topical proparacaine is indicative of centralized neuropathic pain. Changes in pain VAS score reported after proparacaine drop from baseline to 16 weeks will be assessed.
Efficacy of OXERVATE 0.002% at a reduced-dose regime (3 days on/1 day off) in patients reporting ocular side-effects/ocular pain assessed by changes in ocular inflammation on in vivo confocal microscopy. | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  Change in dendritic cell density on in vivo confocal microscopy from baseline to 4 weeks, and at 16 weeks.
Efficacy of OXERVATE 0.002% at an increased-dose regime (6times/daily) for 4 weeks assessed by changes in ocular inflammation on in vivo confocal microscopy. | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  Change in dendritic cell density on in vivo confocal microscopy from baseline and 4 weeks measure, at 8 and 16 weeks.
Changes in aqueous tear production as assessed by Schirmer's II test, change from baseline measurement at 16 weeks. | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  The Schirmer's test will be performed 5 minutes after a drop of topical anesthesia with 0.5% proparacaine (Alcon Inc., Ft Worth TX) is applied to the eye. The Schirmer test is performed by placing a narrow filter-paper strip (5 x 35 mm strip of Whatman #41 filter paper) in the inferior cul-de-sac. The resultant Schirmer strip value will be reported after 5 minutes. Aqueous tear production will be measured by the length in millimeters that the strip wets during 5 minutes. Values less than 10 mm / 5 minutes indicate tear production insufficiency. Values greater than 25 mm / 5 minutes indicate normal tear production as expected from a healthy eye.
Change in the stability of the tear film as assessed by Tear Film Break Up Time (TFBUT), change from baseline measurement at 16 weeks. | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  The standard Tear Break Up Time measurement will be performed by dropping a fluorescein drop to the inferior tarsal conjunctiva and waiting 30 seconds. After several blinks, the tear film will be examined using a broad beam of the slit lamp with a blue filter. The time lapse between the last blink and the appearance of the first randomly distributed dark discontinuity in the fluorescein stained tear film will be measured three times and the mean value of the measurements will be calculated. Break-up times less than 10 seconds are considered abnormal. A positive change from baseline (increase in amount of seconds it take tear film to break up / show discontinuity) indicates improvement.
Changes in ocular surface integrity as assessed by NEI corneal staining scale, changes in corneal fluorescein staining from baseline at 16 weeks. | From Baseline Visit to End of Study Visit (16 weeks post treatment)
  Corneal fluorescein staining will be performed after 2 minutes of application of a fluorescein drop. The entire cornea will be then examined using slit-lamp evaluation with cobalt blue illumination. Staining will be graded using the NEI grading scheme, with a total range of 0-15. Each corneal quadrant (central, superior, temporal, nasal, and inferior) will be graded for severity of staining on a scale of 0-3, 0 being no staining, 1 being mild staining, 2 being moderate staining, and 3 being severe staining. The total of all 5 corneal quadrants will be added together to get the resultant score per eye out of 15. 15/15 represents the most severe staining, whereas 0/15 represents no staining and greater ocular surface integrity and homeostasis.

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No